CLINICAL TRIAL: NCT03207542
Title: An Open-label Phase 2 Trial Evaluating the Efficacy and Safety of Daratumumab in Subjects With Relapsed/Refractory B-cell or T-cell Precursor Acute Lymphoblastic Leukemia (ALL)
Brief Title: Trial Evaluating the Efficacy and Safety of Daratumumab in Subjects With Relapsed/Refractory B-cell or T-cell Precursor Acute Lymphoblastic Leukemia (ALL)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI request
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0973; NCI-2018-01131 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-06-30; First posted 2017-07-02 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Malignant Neoplasms Stated as Primary Lymphoid Haematopoietic
Keywords: Malignant neoplasms stated as primary lymphoid haematopoietic; B-Cell Precursor Acute Lymphoblastic Leukemia; T-Cell Precursor Acute Lymphoblastic Leukemia; ALL; Daratumumab
MeSH Terms: interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- B-Cell Precursor Acute Lymphoblastic Leukemia (ALL) (Experimental): Participants receive Daratumumab by vein over about 4 hours on Days 1, 8, 15, and 22 of Cycles 1 and 2, Days 1 and 15 of Cycles 3-6, and then on Day 1 of Cycles 7 and beyond.
  Each cycle is 28 days.
  Interventions: Drug: Daratumumab
- T-Cell Precursor Acute Lymphoblastic Leukemia (ALL) (Experimental): Participants receive Daratumumab by vein over about 4 hours on Days 1, 8, 15, and 22 of Cycles 1 and 2, Days 1 and 15 of Cycles 3-6, and then on Day 1 of Cycles 7 and beyond.
  Each cycle is 28 days.
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — 16 mg/kg by vein weekly for the first 2 cycles (8 weeks) of treatment, followed by every 2 weeks for 4 cycles (or 16 weeks) and then every 4 weeks until progression or up to 1 year of treatment whichever comes earlier.

SUMMARY:
The goal of this clinical research study is to learn if daratumumab can help to control B- or T-cell acute lymphoblastic leukemia (ALL). The safety of daratumumab will also be studied.

This is an investigational study. Daratumumab is FDA approved and commercially available for treatment of multiple myeloma. It is considered investigational to use daratumumab to treat ALL.

The study doctor can explain how the study drug is designed to work.

Up to 72 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

Each cycle is 28 days.

If you are found to be eligible to take part in this study, you will receive daratumumab by vein over about 4 hours on Days 1, 8, 15, and 22 of Cycles 1 and 2, Days 1 and 15 of Cycles 3-6, and then on Day 1 of Cycles 7 and beyond. Your first dose of daratumumab will be given over about 7 hours.

In this study, the following will be done to lower the chance of a daratumumab infusion related reaction:

* You will get medications, including steroids, acetaminophen, and/or antihistamine before the infusion. If you are considered high risk, you may also get medications, including inhaled steroids, after the infusion.
* The infusion may be slowed down or stopped if you have a reaction.
* You may stay overnight in the hospital after the infusion so the study staff can check your health.

You may ask the study staff for information about how these drugs are given and their risks. You may also be asked to stay in the hospital overnight to watch you for side effects, if needed.

Length of Study:

You may receive daratumumab for up to 1 year. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Study Visits:

Within 24 hours before your first dose of study drug, if you can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

Every 2 weeks during Cycles 1-6, blood (about 1 teaspoon) will be drawn for CMV testing.

On Day 1 of Cycles 1 and 2:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* During Cycle 2, you will have a bone marrow aspirate/biopsy to check the status of the disease.

On Days 8, 15, 22 of Cycles 1 and 2, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 3-6:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* During Cycle 3, you will have an EKG.
* If you can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

On Day 1 of Cycles 3 and beyond, you will have a bone marrow biopsy/aspirate to check the status of the disease. If the disease appears to be responding to the study drug, the study doctor will decide how often you will have this procedure.

On Day 15 of Cycles 3-6, blood (about 2 teaspoons) will be drawn for routine tests.

On Day 1 of Cycles 7 and beyond:

* You will have a physical exam.
* Blood (about 2 teaspoons) will be drawn for routine tests and CMV testing.
* During Cycle 7 only, you will have an EKG.
* If you can become pregnant, blood (about 1 teaspoon) will be drawn for a pregnancy test.

End of Treatment:

About 28-35 days after the last dose of daratumumab:

* You will have a physical exam.
* You will have an EKG.
* Blood (about 2 teaspoons) will be drawn for routine tests.
* If the doctor thinks it is needed, you may have a bone marrow biopsy/aspiration to check the status of the disease.

Follow-Up Visits:

The study staff will call you to ask how you are doing 1 time each month for the first year after your End-of-Treatment visit, then every 6 months during the second year after the visit, and then 1 time every year after that. Each call should last about 5 minutes.

At 30 and 60 days after your last dose of study drug and then every 2-3 months after that for 1 year:

* You will have a physical exam.
* If the disease appeared to be responding to the study drug, blood (about 2 teaspoons) will be drawn for routine tests. Every 4-12 weeks, this sample may be used for CMV testing. If the disease appears to get worse, you will stop having these blood draws.
* If the disease appeared to be responding to the study drug, you will have a bone marrow aspirate and/or biopsy.
* If the disease appeared to be responding to the study drug, you will have an EKG at your first follow-up visit.

After 1 year, you may continue to have follow-up visits as part of your routine care. This will be discussed with you by the study doctor in more detail.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be at least 18 years of age.
2. The subject must have precursor B-cell or T-cell acute lymphoblastic leukemia. B-cell: relapsed or refractory after first or subsequent salvage therapy; or T-cell: relapsed or refractory with first remission duration less than or equal to 12 months in first salvage; or relapsed or refractory after first or subsequent salvage therapy.
3. More than 5% blasts in bone marrow.
4. Eastern Cooperative Oncology Group (ECOG) performance status </= 2.
5. Life expectancy of >/= 12 weeks.
6. Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device, hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin prior to dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy. A man who is sexually active with a woman of childbearing potential must always use a latex or synthetic condom during the study and for 4 months after discontinuing daratumumab.
7. A woman of childbearing potential must have a negative serum or urine pregnancy test at screening within 14 days and again within 72 hours prior to dosing.
8. Each subject must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Subjects must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.

Exclusion Criteria:

1. Active leukemic central nervous system (CNS) disease.
2. Active acute Graft-versus-Host Disease (GvHD) or chronic GVHD grade 2 or higher.
3. Patients who have received prior stem cell transplantation will be allowed to enroll as long as prior transplantation has been at least 3 months before enrollment in the trial and any transplant related toxicities have subsided to Grade 1 or less.
4. Philadelphia chromosome-positive (Ph+) ALL.
5. Cancer chemotherapy within 2 weeks prior to start of daratumumab treatment (steroid or hydroxyurea can be used up to 24 hours prior to first daratumumab infusion for control of high white cell counts)
6. Cancer immunotherapy within four weeks prior to start of daratumumab treatment (exception blinatumomab within two weeks prior)
7. Diagnosed or treated for malignancy other than ALL, except: 1) Malignancy treated with curative intent and with no known active disease present for >/= 3 years before treatment; 2) Adequately treated non-melanoma skin cancer or lentigo maligna or carcinoma in situ (e.g. cervical, breast) without evidence of disease; 3) or malignancy that in the opinion of the investigator, with concurrence with the MDACC IND office, is considered cured with minimal risk of recurrence within 3 years.
8. Subject has known chronic obstructive pulmonary disease (COPD) with a Forced Expiratory Volume in 1 second (FEV1) <50% of predicted normal. NOTE: FEV1 testing is required for patients suspected of having COPD and subjects must be excluded if FEV1 <50% of predicted normal.
9. Subject has known moderate or severe persistent asthma within the past 2 years (see Appendix A: Classification of Asthma Severity), or currently has uncontrolled asthma of any classification. NOTE: subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study.
10. Subject is known to be seropositive for human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibody (unless treated curatively).
11. Subject has any concurrent medical condition or disease (e.g, active systemic infection) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
12. Subject has any of the following laboratory test results at cycle 1 day 1 pre-dosing: 1) Alanine aminotransferase level (ALT) >/= 2.5 x the upper limit of normal (ULN); 2) Aspartate Aminotransferase (AST) >/= 2.5 x the ULN; 3) Total bilirubin level >/= 1.5 x ULN, (except for Gilbert Syndrome: direct bilirubin >/= 1.5 x ULN); 4) Creatinine > 2 x ULN.
13. Subject has clinically significant cardiac disease, including: 1) myocardial infarction within 1 year before study enrollment, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association Class III-IV); 2)uncontrolled cardiac arrhythmia or clinically significant ECG abnormalities; 3) screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
14. Subject has known allergies, hypersensitivity, or intolerance to boron or mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or Investigator's Brochure), or known sensitivity to mammalian-derived products.
15. Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study or within 4 months after the last dose of any component of the treatment regimen. Or, subject is a man who plans to father a child while enrolled in this study or within 4 months after the last dose of any component of the treatment regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) in Participants with Relapsed/Refractory B-Cell or T-Cell Precursor Acute Lymphoblastic Leukemia (ALL) | 12 weeks
  Overall response (OR) defined as achievement of complete remission (CR), CR with only Partial Hematological Recovery (CRp), Complete Response without Hematological Recovery (CRi).
Adverse Events of Daratumumab in Participants with Relapsed/Refractory B-Cell or T-Cell Precursor Acute Lymphoblastic Leukemia (ALL) | 30 days after the last dose of study drug
  Descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.03 utilized for adverse event reporting.

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, MBBS, Principal Investigator — M.D. Anderson Cancer Center

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org